CLINICAL TRIAL: NCT02945228
Title: Drug Use-Results Survey in Patients Infected With Hepatitis C Virus Genotype 2
Brief Title: Drug Use-Results Survey in Participants Infected With Hepatitis C Virus Genotype 2
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-764
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Chronic Hepatitis C Virus
Keywords: Genotype 2; Paritaprevir; Hepatitis C Virus (HCV); Ritonavir; Ombitasvir
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic infection of hepatitis C virus (HCV) genotype 2: Participants with confirmed chronic HCV genotype 2, receiving paritaprevir/ritonavir/ombitasvir and ribavirin according to standard of care and in line with the current local label

SUMMARY:
The main objective of this study is to evaluate the safety and effectiveness of paritaprevir/ritonavir/ombitasvir with ribavirin used for participants infected with chronic hepatitis C virus (HCV) genotype 2 in daily practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

* HCV genotype 2 participants treated with paritaprevir/ritonavir/ombitasvir plus ribavirin in daily practice.

Exclusion Criteria:

* Participants who have been previously treated with paritaprevir/ritonavir/ombitasvir and ribavirin.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Chronic hepatitis C virus (HCV) genotype 2
Sampling Method: Non-Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Sustained Virologic Response (SVR12) | 12 weeks after last dose of study drug.
  Hepatitis C virus (HCV) ribonucleic acid (RNA) less than the lower limit of quantification (LLOQ) 12 weeks after the last dose of study drug.

SECONDARY OUTCOMES:
Percentage of Participants with Virologic Failure During Treatment (breakthrough) | Up to 12 Weeks
  HCV RNA levels reach less than the LLOQ, then increase to greater than or equal to the LLOQ at any point during treatment.
Percentage of Participants with Virologic Failure After Treatment (relapse) | Post-treatment 24 weeks
  Undetectable viremia (HCV RNA less than LLOQ) at the end of the 16 weeks treatment but subsequent viremia (HCV RNA greater than or equal to LLOQ) during the follow-up period of 24 weeks after treatment.
Percentage of Participants with Sustained Virologic Response (SVR24) | 24 weeks after the last dose of study drug
  HCV RNA less than the LLOQ 24 weeks after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (170):
- Japan (170):
  - Aichi Medical University Hosp /ID# 161892, Nagakute, Aichi-ken
  - Matsuyama Red Cross Hosp /ID# 162953, Matsuyama, Ehime
  - NHO Kyushu Medical Center /ID# 162956, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 164158, Kurume-shi, Fukuoka
  - Kusunoki Hospital /ID# 158119, Fujioka, Gunma
  - National Hospital Organization Takasaki General Medical Center /ID# 160877, Takasaki-shi, Gunma
  - NHO Fukuyama Medical Center /ID# 162909, Fukuyama-shi, Hiroshima
  - Fukuyama City Hospital /ID# 161889, Fukuyama-shi, Hiroshima
  - The Hospital of Hyogo College of Medicine /ID# 162913, Nishinomiya-shi, Hyōgo
  - Nanpuh Hospital /ID# 168348, Kagoshima, Kagoshima-ken
  - St. Marianna University School of Medicine Hospital /ID# 160876, Kawasaki, Kanagawa
  - Yokohama City Univ Medical Ctr /ID# 162905, Yokohama, Kanagawa
  - Kumamoto University Hospital /ID# 167048, Kumamoto, Kumamoto
  - Kumamoto Shinto General Hospital /ID# 165275, Kumamoto, Kumamoto
  - Okayama University Hospital /ID# 165268, Okayama, Okayama-ken
  - Osaka Red Cross Hospital /ID# 161888, Osaka, Osaka
  - Osaka City University Hospital /ID# 165290, Osaka, Osaka
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 167688, Osaka, Osaka
  - Osaka Medical College Hospital /ID# 162908, Takatsuki -shi, Osaka
  - Saitama Medical Center, Saitama Medical University /ID# 162911, Kawagoe-shi, Saitama
  - Dokkyo Medical University Saitama Medical Center /ID# 162907, Koshigaya, Saitama
  - Hamamatsu University Hospital /ID# 171048, Hamamatsu, Shizuoka
  - Tokyo Jikei Daisan Hospital /ID# 164159, Komae-shi, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 167685, Shinjuku-ku, Tokyo
  - University of Yamanashi Hospital /ID# 161770, Chuo-shi, Yamanashi
  - Kato Michio Hepatology Clinic /ID# 159476, Amagasaki, Hyogo
  - Aomori Prefectural Central Hos /ID# 160822, Aomori
  - Mantani Clinic /ID# 168353, Arida
  - Japanese Red Cross Asahikawa /ID# 165265, Asahikawa
  - Asahikawa City Hospital /ID# 167703, Asahikawa-shi
  - National Hospital Organization /ID# 168346, Chiba
  - Chiba University Hospital /ID# 160875, Chiba
  - Seirei Sakura Citizen Hospital /ID# 166896, Chiba
  - Kenseido-iin /ID# 164166, Chichibu
  - Fuji City General Hospital /ID# 165278, Fuji
  - Fukui Prefectural Hospital /ID# 168344, Fukui
  - Fukui Prefectural Hospital /ID# 169552, Fukui
  - University of Fukui Hospital /ID# 166933, Fukui
  - Chihaya Hospital /ID# 161893, Fukuoka
  - Morichika Internal Medicine /ID# 168351, Fukuyama
  - Gifu Municipal Hospital /ID# 165287, Gifu
  - Shiroyama Hospital /ID# 164963, Habikino-osaka
  - Aomori Rosai Hospital /ID# 167702, Hachinohe
  - Tamakoshi Clinic /ID# 165282, Hamamatsu
  - Higashihiroshima Medical Ctr /ID# 168343, Higashihiroshima
  - Mito Medical Center /ID# 171046, Higashiibaraki-gun
  - Higashiomicity Notogawa Hosp /ID# 161891, Higashiomi, Shiga
  - Shin-ishikiri Clinic /ID# 169643, Higashiosaka
  - Wakakusa Daiichi Hospital /ID# 166882, Higashiosaka
  - Hiroshima Red Cross Hosp Atomi /ID# 162912, Hiroshima
  - Hiroshima University Hospital /ID# 160815, Hiroshima
  - Hiroshima-Nishi Medical Center /ID# 169642, Hiroshima
  - Koyo New Town Hospital /ID# 161890, Hiroshima
  - Taishi Hospital /ID# 165291, Hyōgo
  - Iizuka Hospital /ID# 161886, Iizuka
  - Ikeda Municipal Hospital /ID# 160814, Ikeda
  - Tokyo Med Uni Ibaraki Med Ctr /ID# 162955, Inashiki
  - Nippon Med Chiba Hokusoh Hosp /ID# 162902, Inzai
  - Saitama Medical University Hos /ID# 161768, Iruma-gun
  - Itoigawa Sogo Hospital /ID# 166884, Itoigawa
  - Kamiiwade Internal Med-Neuro /ID# 166881, Iwade
  - Kaizuka City Hospital /ID# 165256, Kaizuka
  - Kamisu Saiseikai Hospital /ID# 167701, Kamisu
  - Kiyokawa Hospital /ID# 164961, Kanagawa
  - Hiratsuka City Hospital /ID# 161884, Kanagawa
  - Niwa Hospital /ID# 167684, Kanagawa
  - Fuji Clinic /ID# 160820, Kan’onjichō
  - Ibaraki Prefectural Cent. Hosp /ID# 164962, Kasama
  - The Jikei Univ. Kashiwa Hosp. /ID# 166888, Kashiwa-shi
  - Kashiwazaki General Hospital a /ID# 168352, Kashiwazaki
  - Kawase Clinic /ID# 164957, Kasugai
  - Hirose Clinic /ID# 167699, Kawagoe
  - Sekishindo Hospital /ID# 162960, Kawagoe
  - Kawaguchi Municipal Medical Ce /ID# 165270, Kawaguchi
  - Kawasaki Municipal Tama Hospit /ID# 165267, Kawasaki
  - Kanto Rosai Hospital /ID# 165258, Kawasaki-shi, Kanagawa
  - Kishiwada Tokushukai Hospital /ID# 164964, Kishiwada, Osaka
  - Kokura Kinen Hospital /ID# 164969, Kitakyushu
  - Kitasato University Medical Ce /ID# 158120, Kitamoto
  - Kobe Asahi Hospital /ID# 161896, Kobe
  - Kobe Adventist Hospital /ID# 161897, Kobe
  - Konan Kosei Hospital /ID# 165277, Konan-shi
  - Hanada Internal Medicine Clin /ID# 165266, Koshigaya, Saitam
  - Cosmos Clinic /ID# 164161, Kōriyama
  - Ishida Medical Clinic /ID# 166887, Kōriyama
  - Kawasaki Medical School Hosp /ID# 162906, Kurashiki
  - National Hosp Org Kure Med Cen /ID# 167689, Kure, Hiroshima
  - Kurihara Central Hospital /ID# 171047, Kurihara
  - Kuroishi Hospital /ID# 164971, Kuroishi-aomori
  - Shin Koga Clinic /ID# 164972, Kurume
  - Koga Hospital 21 /ID# 167698, Kurume
  - Hori Internal Medicine Clinic /ID# 167696, Kushiro
  - NHO Kyoto Medical Center /ID# 162910, Kyoto
  - Matsuzaki Internal Medicine Cl /ID# 164970, Kyoto
  - Gibo Hepatorogy Clinic /ID# 161766, Matsumoto
  - Kizawa Memorial Hospital /ID# 162957, Minokamo
  - Sumiyoshi Clinic Hospital /ID# 164163, Mito
  - South Miyagi Medical Center /ID# 164965, Miyagi
  - National Hospital Organization /ID# 168345, Miyakonojō
  - Miyazaki Medical Center Hospit /ID# 165279, Miyazaki
  - University of Miyazaki Hosp /ID# 166880, Miyazaki
  - Matsushita Memorial Hospital /ID# 167693, Moriguchi-shi
  - Suzuki Clinic /ID# 165264, Nagareyama
  - Meitetsu Hospital /ID# 165288, Nagoya
  - Nagoya Central Hospital /ID# 166879, Nagoya
  - Aikawa Minnano-shinryojo /ID# 164168, Nagoya
  - Meijo Hospital /ID# 164966, Nagoya-aichi
  - Nara City Hospital /ID# 162959, Nara
  - Tani Internal Medicine Clinic /ID# 164974, Nayoro
  - Ooka Clinic /ID# 161887, Nishinomiya
  - Noshiro Yamamoto Med. Assoc. /ID# 162964, Noshiro
  - Manna Clinic /ID# 169548, Odawara
  - Okayama Saiseikai Outpatient Center Hospital /ID# 159475, Okayama
  - Omuta City Hospital /ID# 164967, Omuta
  - Kita-harima Medical Center /ID# 164165, Ono
  - Onomichi Central General Hospi /ID# 162903, Onomichi
  - Kenporen Osaka Central Hospita /ID# 164956, Osaka
  - Asai Naika /ID# 167691, Osaka
  - Osaka Inter. Cancer Institute /ID# 166889, Osaka
  - Osaka Police Hospital /ID# 161769, Osaka
  - Asai Naika Iin /ID# 164955, Osaka
  - Utajima Ueda Clinic /ID# 161894, Osaka
  - Tamai Clinic /ID# 164162, Osaka
  - Osaka Hospital /ID# 164157, Osaka
  - Oita Midical Center /ID# 164960, Ōita
  - Seko Internal Medicine Clinic /ID# 164169, Ōtsu
  - Kawazoe Internal Medicine Clin /ID# 165292, Saga
  - Saitama Citizens Medical Ctr /ID# 169550, Saitama
  - Sainokuni Higashiomiya Medical /ID# 167700, Saitama
  - Honda Internal Clinic /ID# 161767, Saitama
  - Saitama Cooperative Hospital /ID# 167697, Saitama
  - Minamitani Clinic /ID# 160821, Sakai
  - Kaisei Hospital /ID# 164973, Sapporo
  - Sendai Kousei Hospital /ID# 162961, Sendai
  - Saka General Hospital /ID# 162962, Shiogama-miyagi
  - Saiseikai Suita Hospital /ID# 165289, Suita
  - Suita Municipal Hospital /ID# 164958, Suita-osaka
  - Kagawa Prefectural Central Hos /ID# 160816, Takamatsu
  - Sawada Hepatology & Gastro /ID# 165255, Takaraduka
  - Tenjin Tanaka Internal Medicin /ID# 166883, Takatsuki
  - Hamada Clinic /ID# 171045, Tatebayashi
  - Todachuo General Hospital /ID# 165280, Toda-shi, Saitama
  - Eastern Chiba Medical Center /ID# 165257, Togane, Chiba
  - Delta Clinic /ID# 164167, Tokorozawa
  - The Jikei University Hospital /ID# 169547, Tokyo
  - Abbott Japan /ID# 144983, Tokyo
  - Juntendo University Hospital /ID# 161771, Tokyo
  - Nippon Medical School Hospital /ID# 164164, Tokyo
  - Tokyo Metropolitan Bokutoh Hos /ID# 167686, Tokyo
  - Ohashi Medical Office /ID# 164968, Tokyo
  - Juntendo Univ Nerima Hosp /ID# 164160, Tokyo
  - JP Red Cross Musashino Hosp /ID# 162904, Tokyo
  - Toyama University Hospital /ID# 169551, Toyoma
  - Toyonaka Municipal Hospital /ID# 167692, Toyonaka
  - Ehime University Hospital /ID# 161885, Tōon
  - Mie Syokaki Clinic /ID# 161895, TSU, MIE
  - Saiseikai Utsunomiya Hospital /ID# 162958, Utsunomiya
  - Seike Clinic /ID# 166890, Uwajima
  - Saiseikai Wakayama Hospital /ID# 162954, Wakayama
  - Wakayama Rosai Hospital /ID# 165254, Wakayama
  - Tokyo Women's Medical Universi /ID# 167694, Yachiyo
  - Tohoku Central Hospital /ID# 166897, Yamagata
  - Okuda Gastrointestinal Medicin /ID# 168349, Yamaguchi
  - Kainan Hospital /ID# 164959, Yatomi-shi
  - Kumamoto Rosai Hospital /ID# 167695, Yatsushiro-shi
  - Mie Prefectural General Medica /ID# 162963, Yokkaichi
  - Showa Univ Fujigaoka Hosp /ID# 162952, Yokohama
  - Oita University Hospital /ID# 169549, Yufu-shi
  - Yamaguchi Surgery Clinic /ID# 167704, Yugawara
  - Josai Hospital /ID# 168347, Yūki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/ombitasvir_P15-764.pdf